CLINICAL TRIAL: NCT01340690
Title: PAD-study: Nutritional Efficacy of Polyunsaturated Fatty Acids (Omega-3 and Omega-6) in Combination With Zinc and Magnesium Versus Placebo in Children and Adolescents With Attention Deficit/ Hyperactivity Disorder (ADHD)
Brief Title: Efficacy Study of Polyunsaturated Fatty Acids in Children and Adolescents With Attention Deficit/ Hyperactivity Disorder
Acronym: PAD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sample size of the planned interims analysis was achieved
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Engelhard Arzneimittel GmbH & Co.KG (Industry)
Responsible Party: Principal Investigator, Prof. Huss, Michael Huss, Prof. Dr., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAD-EA-10-01-067
Record Dates: First submitted 2011-04-07; First posted 2011-04-22 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: ADHD
Keywords: ADHD; children; adolescents; Polyunsaturated Fatty Acids; ADHDRS - IV
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Suspensions

STUDY DESIGN:
Intervention Model Description: We use the dietary supplementation like a medication and performed the study like a phase 3 medication study, because the dietary supplementation (verum) is available as special preparation in drug stores.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The verum "nutrional supplementation" is completely masked and an appropriate Placebo is provided. Up to know, none of the above mentioned is unblinded
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ω-3 fatty acids suspension (Active Comparator): 2 bags of Esprico(R) suspension each day. Each 4ml suspension bag includes 400mg eicosapentaenoic acid (EPA), 40mg docosahexaenoic acid (DHA), 5.4 mg gamma-linolenic acid (GLA), 80 mg magnesium, 5 mg zinc and consists of linseed oil, xylitol, sea fish oil with high portion of omega-3-acids, magnesium citrate, vegetable oil, orange flavour, evening primrose oil, zink gluconate, soya lecithin, citric acid, acesulfame k (E950)
  Interventions: Dietary Supplement: ω-3 fatty acids suspension
- placebo suspension (Placebo Comparator): 2 bags of Esprico (R) placebo suspension. Includes no ω-3 fatty acids, no ω-6 fatty acids, no magnesium and no zinc, but other vegetable oils, orange flavor, etc.
  Interventions: Dietary Supplement: placebo suspension

INTERVENTIONS:
Dietary Supplement: ω-3 fatty acids suspension — 2 bags of Esprico(R) suspension given orally once daily in the morning for 84 days
  Other Names: Esprico(R) suspension; 2 verum to 1 placebo
  Arms: ω-3 fatty acids suspension
Dietary Supplement: placebo suspension — suspension to mimic verum Esprico (R) suspension. 2 bags of Esprico(R) placebo suspension given orally once daily in the morning for 84 days
  Arms: placebo suspension

SUMMARY:
This study will determine the nutritional efficacy of Polyunsaturated Fatty Acids (PUFAs) in combination with zinc and magnesium, in children and adolescents diagnosed with Attention Deficit/ Hyperactivity Disorder (ADHD). The nutritional efficacy has to be proven in agreement with the German "Verordnung über Diätetische Lebensmittel (DiätV)" and the corresponding European Directive 1999/21/EC. This objective is reached by performing a placebo-controlled supplementation study with a main efficacy criterion which is also being used in pivotal studies of stimulant and non-stimulant drugs, i.e. the treatment differences between final visit and baseline in the Attention Deficit Hyperactivity Disorder Rating Scale, Parent Version IV (ADHDRS-IV).

DETAILED DESCRIPTION:
The syndrome of ADHD affects 5-6% of the children and adolescents worldwide. The hallmarks are inattention, impulsivity and hyperactivity. Due to parent's fear of significant adverse effects caused by stimulant or non-stimulant therapy a high degree of children with ADHD remains untreated. Recent observational studies showed that ADHD is often associated with decreased nutritional status of certain PUFAs, zinc and magnesium which might be due to metabolic disturbances in the case of fatty acids. First interventional studies revealed that a supplementation of these nutrients may affect ADHD-related disorders and might improve certain clinical parameters, such as concentration.

Participants will be randomly assigned to receive either a nutritional supplement or placebo once a day for the duration of 84 days. Participants will come in for the assessment of ADHD symptoms, compliance and the assessment of secondary outcome variables. Side effects will be monitored continuously and also assessed by rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent by parents and patients (separately for age groups 6 - 11 years and 12 - 17 years)
* Children and adolescents of both gender in the age group between 6 and 17 years
* Confirmed diagnosis of ADHD by semi-structured clinical interview Kiddie Schedule for Affective Disorders and Schizophrenia for school-age children (K-SADS)
* ADHDRS-IV-Parent Version (18-Item-Scale): Investigator Administered and Scored ≥24
* Sufficient knowledge of the German language

Exclusion Criteria:

* Known hypersensitivity against components of either the verum or placebo food
* All serious internal diseases
* All severe psychiatric diseases except oppositional defiant disorders
* Current intake of the following medication: antidepressants and other psychotropic medication
* Recent intake of ω-3 fatty acids supplementation
* Indication for hospitalization
* Suicidality (including suicidal thoughts)
* intelligence quotient < 70
* Previous medication with stimulants within 4 weeks
* Placement in an institution on official or judicial ruling
* Lack of willingness to store and transmit pseudonym data according to German regulations
* Parallel participation in another trial, or less than 4 weeks ago
* Patients foreseeable requiring a primary medication with methylphenidate during the study period of 12 weeks

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2011-03-08 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
ADHDRS - IV | Difference in total score between baseline and end of study, an expected average of 84 days
  The primary outcome measure for efficacy will be the absolute change in the ADHDRS total score between baseline and day 84 of randomized treatment.

SECONDARY OUTCOMES:
Barkley´s Side Effects Rating Scale | Baseline and each visit, monthly, an expected average of 84 days in total
  Number of Participants with Adverse Events.
Montgomery-Åsberg-Depression Rating Scale (MADRS) | Baseline and each visit, monthly, an expected average of 84 days in total
  Assessment of Symptoms of Depression.
Continuous Performance Test (CPT) | change from Baseline to end of treatment, an expected average of 84 days
  Differences in Continuous Performance Test.
Nutrition protocol | baseline
  Assessment of diet habits.
Weiss Functional Impairment Rating Scale - Parent Report (WFIRS-P) | change from Baseline to end of treatment, an expected average of 84 days
  Assessment of Symptoms of ADHD and to what degree individual's behavior or emotional problems have impacted various clinically relevant domains of functioning.
PUFA associated blood parameters | change from Baseline to end of treatment, an expected average of 84 days
  complete fatty acid profile in red blood cells and relevant ratios, e.g. Omega-HS-Index, Plasma-Zinc, Plasma-Copper, Serum-Magnesium, Serum-Ferritin,...

CONTACTS AND LOCATIONS:
Overall Officials: Michael Huss, Prof. Dr., Principal Investigator — University Medicine, Mainz, Dep. of Child and Adolescent Psychiatry
Locations (5):
- Germany (5):
  - DRK Fachklinik für Kinder- und Jugendpsychiatrie, Psychotherapie, Psychosomatik, Bad Neuenahr
  - Charité - Universitätsmedizin Berlin, CVK Klinik für Psychiatrie, Psychosomatik und Psychotherapie des Kindes- und Jugendalters, Berlin
  - University Medicine Mainz, Mainz
  - Kinderzentrum Maulbronn gGmbH, Maulbronn
  - Johanniter - Zentrum für Kinder- und Jugendpsychiatrie Neuwied, Neuwied

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schuchardt JP, Huss M, Stauss-Grabo M, Hahn A. Significance of long-chain polyunsaturated fatty acids (PUFAs) for the development and behaviour of children. Eur J Pediatr. 2010 Feb;169(2):149-64. doi: 10.1007/s00431-009-1035-8. Epub 2009 Aug 12. PMID 19672626
- [Background] Huss M, Volp A, Stauss-Grabo M. Supplementation of polyunsaturated fatty acids, magnesium and zinc in children seeking medical advice for attention-deficit/hyperactivity problems - an observational cohort study. Lipids Health Dis. 2010 Sep 24;9:105. doi: 10.1186/1476-511X-9-105. PMID 20868469